CLINICAL TRIAL: NCT01602380
Title: A Randomised, Double-blind, Parallel-group, Multicentre, Phase III Study to Compare the Efficacy and Tolerability of Fulvestrant (FASLODEX) 500 mg With Anastrozole (ARIMIDEX) 1 mg as Hormonal Treatment for Postmenopausal Women With Hormone Receptor-Positive Locally Advanced or Metastatic Breast Cancer Who Have Not Previously Been Treated With Any Hormonal Therapy.
Brief Title: A Global Study to Compare the Effects of Fulvestrant and Arimidex in a Subset of Patients With Breast Cancer.
Acronym: FALCON
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D699BC00001; 2011-006326-24 (EudraCT Number)
Record Dates: First submitted 2012-05-11; First posted 2012-05-21 (Estimated); Results first posted 2017-05-17 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Hormone Receptor Positive Breast Cancer
Keywords: hormone receptor positive breast cancer; endocrine; no hormone therapy; hormone; breast; cancer; neoplasm; metastatic; tumour
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis | interventions — Fulvestrant; Anastrozole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- faslodex+placebo (Experimental): Blinded: Fulvestrant 500mg intramuscular injection (2x250mg) plus dummy Anastrozole tablets
  Interventions: Drug: faslodex 500mg; Drug: arimidex dummy
- arimidex +placebo (Active Comparator): Blinded: Anastrozole 1mg tablets plus dummy Fulvestrant intramuscular injection (2x0mg)
  Interventions: Drug: arimidex 1mg; Drug: faslodex dummy

INTERVENTIONS:
Drug: faslodex 500mg — 2 x intramuscular injections at day 1, 14, 28 and every 28 days thereafter
  Arms: faslodex+placebo
Drug: arimidex 1mg — oral tablet 1 daily
  Arms: arimidex +placebo
Drug: faslodex dummy — 2 x intramuscular injections at day 1, 14, 28 and every 28 days thereafter
  Arms: arimidex +placebo
Drug: arimidex dummy — oral tablet 1 daily
  Arms: faslodex+placebo

SUMMARY:
The purpose of the study is to compare how treatment with Fulvestrant (FASLODEX) or Anastrozole (ARIMIDEX) effects disease progression for women with locally advanced or metastatic breast cancer who have not had prior hormonal treatment.

DETAILED DESCRIPTION:
A Randomised, Double-blind, Parallel-group, Multicentre, Phase III Study to Compare the Efficacy and Tolerability of Fulvestrant (FASLODEX) 500 mg with Anastrozole (ARIMIDEX) 1 mg as Hormonal Treatment for Postmenopausal Women with Hormone Receptor-Positive Locally Advanced or Metastatic Breast Cancer Who Have Not Previously Been Treated With Any Hormonal Therapy.

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmation of breast cancer in post menopausal women (age >=60). Positive hormone receptor status (ER +ve and/or PgR +ve) of primary or metastatic tumour tissue based on local laboratory assessment.
* EITHER locally advanced disease (1 line of chemotherapy allowed only if remain unsuitable for therapy of curative intent) OR Metastatic disease. (1 line of chemotherapy for breast cancer allowed only if subsequent evidence of further progressive disease)
* At least 1 lesion (measurable and/or non-measurable) that can be accurately assessed at baseline and is suitable for repeated assessment.
* Postmenopausal women, fulfilling 1 of:

  * Prior bilateral oophorectomy
  * Age >60 years
  * Age < 60 years and amenorrheic for 12+months in the absence of chemotherapy, tamoxifen, toremifene, or ovarian suppression and FSH and oestradiol in the postmenopausal range

Exclusion Criteria:

* Presence of life-threatening metastatic disease
* Any of:

  * Extensive hepatic involvement
  * involving brain or meninges
  * symptomatic pulmonary lymph spread
* Discrete lung metastases are acceptable if respiratory function is not significantly compromised
* Prior systemic therapy for breast cancer other than one line of cytotoxic chemotherapy (the last dose of chemotherapy must have been received more than 28 days prior to randomisation)
* Radiation therapy if not completed within 28 days prior to randomisation (with the exception of radiotherapy given for control of bone pain, started prior to randomisation). Prior hormonal treatment for breast cancer.
* Current or prior malignancy within previous 3 years (other than breast cancer or adequately treated basal cell or squamous cell carcinoma of the skin or in situ carcinoma of the cervix).

Ages: 18 Years to 130 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 462 (Actual)
Dates: Start 2012-10-17 (Actual); Primary Completion 2016-04-11 (Actual); Study Completion 2027-08-06 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Shankar S, MD, Study Director — AstraZeneca; John Robertson, MD, Principal Investigator — Graduate Medicine and Health School, University of Nottingham, UK; Matthew Ellis, DM, Principal Investigator — Washington University School of Medicine, USA
Locations (97):
- United States (12):
  - Research Site, Modesto, California
  - Research Site, Savannah, Georgia
  - Research Site, Auburn, Maine
  - Research Site, Worcester, Massachusetts
  - Research Site, Detroit, Michigan
  - Research Site, St Louis, Missouri
  - Research Site, Lincoln, Nebraska
  - Research Site, Somerset, New Jersey
  - Research Site, Columbus, Ohio
  - Research Site, Montgomery, Ohio
  - Research Site, Memphis, Tennessee
  - Research Site, Salt Lake City, Utah
- Argentina (4):
  - Research Site, La Rioja
  - Research Site, Mar del Plata
  - Research Site, Pergamino
  - Research Site, Rosario
- Brazil (2):
  - Research Site, Porto Alegre
  - Research Site, Santo André
- Canada (5):
  - Research Site, Abbotsford, British Columbia
  - Research Site, Vancouver, British Columbia
  - Research Site, Kitchener, Ontario
  - Research Site, Thunder Bay, Ontario
  - Research Site, Montreal, Quebec
- China (8):
  - Research Site, Chengdu
  - Research Site, Dalian
  - Research Site, Fuzhou
  - Research Site, Guangzhou
  - Research Site, Shanghai
  - Research Site, Shenyang
  - Research Site, Suzhou
  - Research Site, Tianjin
- Czechia (2):
  - Research Site, Prague
  - Research Site, Příbram
- Italy (8):
  - Research Site, Avellino
  - Research Site, Bari
  - Research Site, Benevento
  - Research Site, Catania
  - Research Site, Genova
  - Research Site, Pisa
  - Research Site, Roma
  - Research Site, Treviglio
- Japan (10):
  - Research Site, Fukuoka
  - Research Site, Hamamatsu
  - Research Site, Kagoshima
  - Research Site, Kumamoto
  - Research Site, Matsuyama
  - Research Site, Mitaka-shi
  - Research Site, Nishinomiya-shi
  - Research Site, Osaka
  - Research Site, Sakaishi
  - Research Site, Suita-shi
- Mexico (3):
  - Research Site, Mexico City
  - Research Site, Mérida
  - Research Site, Monterrey
- Research Site, Lima, Peru
- Poland (3):
  - Research Site, Katowice
  - Research Site, Lodz
  - Research Site, Lublin
- Romania (4):
  - Research Site, Brăila
  - Research Site, Craiova
  - Research Site, Onești
  - Research Site, Timișoara
- Russia (6):
  - Research Site, Barnaul
  - Research Site, Moscow
  - Research Site, Omsk
  - Research Site, Ryazan
  - Research Site, Saint Petersburg
  - Research Site, Tomsk
- Slovakia (3):
  - Research Site, Bardejov
  - Research Site, Bratislava
  - Research Site, Trenčín
- South Africa (3):
  - Research Site, Cape Town
  - Research Site, Pietermaritzburg
  - Research Site, Pretoria
- Spain (6):
  - Research Site, Madrid
  - Research Site, Pamplona
  - Research Site, Pozuelo de Alarcón
  - Research Site, Sabadell
  - Research Site, Seville
  - Research Site, Valencia
- Taiwan (2):
  - Research Site, Taichung
  - Research Site, Taipei
- Turkey (Türkiye) (2):
  - Research Site, Ankara
  - Research Site, Gaziantep
- Ukraine (10):
  - Research Site, Cherkasy
  - Research Site, Dnipro
  - Research Site, Donetsk
  - Research Site, Ivano-Frankivsk
  - Research Site, Kharkiv Region
  - Research Site, Kyiv
  - Research Site, Lviv
  - Research Site, Mariupol
  - Research Site, Uzhhorod
  - Research Site, Vinnytsia
- United Kingdom (3):
  - Research Site, Airdrie
  - Research Site, Derby
  - Research Site, Stoke-on-Trent

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Robertson JFR, Shao Z, Noguchi S, Bondarenko I, Panasci L, Singh S, Subramaniam S, Ellis MJ. Fulvestrant Versus Anastrozole in Endocrine Therapy-Naive Women With Hormone Receptor-Positive Advanced Breast Cancer: Final Overall Survival in the Phase III FALCON Trial. J Clin Oncol. 2025 May;43(13):1539-1545. doi: 10.1200/JCO.24.00994. Epub 2025 Jan 7. PMID 39772884
- [Derived] Robertson JFR, Cheung KL, Noguchi S, Shao Z, Degboe A, Lichfield J, Thirlwell J, Fazal M, Ellis MJ. Health-related quality of life from the FALCON phase III randomised trial of fulvestrant 500 mg versus anastrozole for hormone receptor-positive advanced breast cancer. Eur J Cancer. 2018 May;94:206-215. doi: 10.1016/j.ejca.2018.02.026. Epub 2018 Mar 22. PMID 29574365
- [Derived] Robertson JFR, Bondarenko IM, Trishkina E, Dvorkin M, Panasci L, Manikhas A, Shparyk Y, Cardona-Huerta S, Cheung KL, Philco-Salas MJ, Ruiz-Borrego M, Shao Z, Noguchi S, Rowbottom J, Stuart M, Grinsted LM, Fazal M, Ellis MJ. Fulvestrant 500 mg versus anastrozole 1 mg for hormone receptor-positive advanced breast cancer (FALCON): an international, randomised, double-blind, phase 3 trial. Lancet. 2016 Dec 17;388(10063):2997-3005. doi: 10.1016/S0140-6736(16)32389-3. Epub 2016 Nov 29. PMID 27908454
- [Derived] Ellis MJ, Llombart-Cussac A, Feltl D, Dewar JA, Jasiowka M, Hewson N, Rukazenkov Y, Robertson JF. Fulvestrant 500 mg Versus Anastrozole 1 mg for the First-Line Treatment of Advanced Breast Cancer: Overall Survival Analysis From the Phase II FIRST Study. J Clin Oncol. 2015 Nov 10;33(32):3781-7. doi: 10.1200/JCO.2015.61.5831. Epub 2015 Sep 14. PMID 26371134
- See also: CSP redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D699BC00001&attachmentIdentifier=3c5fd923-5864-4f78-a758-2711d63dd8cd&fileName=D699BC00001-CSP-V6_Redacted_PDFA.pdf&versionIdentifier=
- See also: SAP redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D699BC00001&attachmentIdentifier=09996f70-c58c-4069-a4e4-ab16ccbdf425&fileName=D699BC00001-SAP-Addendum-Edition-2_Redacted_PDFA.pdf&versionIdentifier=
- See also: CSR Synopsis redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D699BC00001&attachmentIdentifier=4dceef94-df4d-490a-aace-7cd49d7f9038&fileName=D699BC00001_CSR_Synopsis_Redacted_PDFA.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient enrolled: 17 October 2012.
Pre-assignment Details: 524 patients were enrolled (signed informed consent). Patients were assigned to treatment if they met all inclusion and none of the exclusion criteria. 62 patients were not randomised, mainly due to eligibility criteria not being fulfilled (44/62 patients) or patient decision (13/62 patients). 462 patients were randomised to receive treatment.
Groups:
- Fulvestrant 500 mg: Patients received fulvestrant (Faslodex™) 500 milligrams (mg), administered as two 5 milliliters (mL) intramuscular injections, 1 in each buttock, at each visit on Days 0, 14 (±3), 28 (±3) and every 28 (±3) days thereafter. In order to support the double-blind, double-dummy design of the trial, each patient randomised to receive fulvestrant, also received placebo to match the anastrozole schedule (tablets, once daily).
- Anastrozole 1 mg: Patients received anastrozole (Arimidex™), administered orally as a single tablet at a dose of 1 mg/day from randomisation on Day 0 and once daily thereafter. In order to support the double-blind, double-dummy design of the trial, each patient randomised to receive anastrozole also received placebo to match the fulvestrant schedule (injections on Days 0, 14 [±3], 28 [±3] and every 28 [±3] days thereafter).
Period: Overall Study
Arm/Group | Fulvestrant 500 mg | Anastrozole 1 mg
Started | 230 | 232
Completed | 25 | 31
Not Completed | 205 | 201
Not completed — Death | 147 | 145
Not completed — Withdrawal by Subject | 39 | 41
Not completed — Lost to Follow-up | 15 | 12
Not completed — Eligibility criteria not fulfilled | 2 | 3
Not completed — Other | 2 | 0

BASELINE CHARACTERISTICS:
Population: The intention to treat (ITT) analysis set included all randomised patients.
Groups:
- Fulvestrant 500 mg: Patients received fulvestrant (Faslodex™) 500 mg, administered as two 5 mL intramuscular injections, 1 in each buttock, at each visit on Days 0, 14 (±3), 28 (±3) and every 28 (±3) days thereafter. In order to support the double-blind, double-dummy design of the trial, each patient randomised to receive fulvestrant, also received placebo to match the anastrozole schedule (tablets, once daily).
- Total: Total of all reporting groups
Arm/Group | Fulvestrant 500 mg | Anastrozole 1 mg | Total
Number analyzed (Participants) | 230 | 232 | 462
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.8 (9.86) [38 to 87] | 63.3 (10.38) [36 to 90] | 63.5 (10.12) [36 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 230 | 232 | 462
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 5 | 6
  Asian | 36 | 34 | 70
  Black or African American | 4 | 4 | 8
  White | 175 | 174 | 349
  Other | 14 | 15 | 29

OUTCOME MEASURES:

1. Primary Outcome: Comparison of Progression-Free Survival (PFS) in Patients Treated With Fulvestrant With Those Treated With Anastrozole
Description: PFS was defined as the time from randomisation until objective disease progression according to Response Evaluation Criteria in Solid Tumours version 1.1 (RECIST 1.1), surgery or radiotherapy to manage worsening of disease or death by any cause (in the absence of progression). Outcome measure is reported as median time from randomisation to PFS, calculated using the Kaplan-Meier technique.
Time Frame: Baseline RECIST 1.1 assessments (Day 0) and then every 12 weeks until the earliest of disease progression evident, patient dies or has surgery/radiotherapy for their disease (up to approximately 38 months)
Population: The ITT analysis set included all randomised patients.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Fulvestrant 500 mg | Anastrozole 1 mg
Number analyzed (Participants) | 230 | 232
Months | 16.6 [13.83 to 20.99] | 13.8 [11.99 to 16.59]
Statistical Analysis 1: Comparison: Fulvestrant 500 mg vs Anastrozole 1 mg; If the true PFS HR for comparison of fulvestrant vs. anastrozole was 0.69 (likely to correspond to a 45% prolongation of PFS) the study had 90% power to demonstrate a statistically significant difference for PFS with a one-sided type 1 error of 2.5% (two-sided 5%); Test type: Superiority or Other; p = 0.0486, Log Rank — 2-sided p-value; Stratified log-rank test with factors for prior chemotherapy for locally advanced or metastatic disease and measurable disease at baseline; Hazard Ratio (HR) = 0.797, 95% CI 2-sided [0.637 to 0.999] — A hazard ratio < 1 favours fulvestrant

2. Secondary Outcome: Comparison of Overall Survival (OS) in Patients Treated With Fulvestrant With Those Treated With Anastrozole; Percentage of Patients With Events
Description: OS was defined as the time from randomisation until death by any cause. The current OS data correspond to that of the final analysis and the outcome measure is reported as percentage of patients with events.
Time Frame: Baseline (Day 0) up to data cut-off for final analysis (up to approximately 116 months). Following disease progression, patients were to be contacted at 12 weekly intervals to determine survival status
Population: The ITT analysis set included all randomised patients. Date of death of 2 participants were unknown in the Anastrozole 1mg arm, hence they were censored for OS analysis.
Measure: Number; unit: Percentage of patients
Arm/Group | Fulvestrant 500 mg | Anastrozole 1 mg
Number analyzed (Participants) | 230 | 232
Percentage of patients | 68.3 | 67.7
Statistical Analysis 1: Comparison: Fulvestrant 500 mg vs Anastrozole 1 mg; 65% OS maturity; Test type: Superiority or Other; p = 0.7579, Log Rank — 2-sided p-value; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.966, 95% CI 2-sided [0.773 to 1.206] — A HR of <1 favours fulvestrant

3. Secondary Outcome: Objective Response Rate (ORR) for Fulvestrant Treatment Versus Anastrozole Treatment
Description: ORR was defined as the percentage patients with an objective response (i.e. those recording a partial response [PR] or complete response [CR]) at some point during the study, prior to disease progression. ORR was assessed in patients with measurable disease at baseline only. The determination of measurable disease at baseline was done using baseline RECIST data. CR was disappearance of all target lesions since baseline; was any pathological lymph nodes selected as target lesions (TL) to have a reduction in short axis to <10 millimeter. PR was at least a 30% decrease in the sum of the diameters of TL, taking as reference the baseline sum of diameters.
Time Frame: Baseline RECIST 1.1 assessments (Day 0) and then every 12 weeks until disease progression or treatment discontinuation (up to approximately 38 months)
Population: Percentages for ORR were calculated based on the number of patients in the ITT analysis set (which included all randomised patients) who had measurable disease at baseline (n=193 for Fulvestrant arm and n=196 for Anastrozole arm).
Measure: Number; unit: Percentage of participants
Arm/Group | Fulvestrant 500 mg | Anastrozole 1 mg
Number analyzed (Participants) | 193 | 196
Percentage of participants | 46.1 | 44.9
Statistical Analysis 1: Comparison: Fulvestrant 500 mg vs Anastrozole 1 mg; Test type: Superiority or Other; p = 0.7290, Regression, Logistic — 2-sided p-value; Odds Ratio (OR) = 1.074, 95% CI 2-sided [0.716 to 1.614]

4. Secondary Outcome: Duration of Response (DoR) for Fulvestrant Treatment Versus Anastrozole Treatment
Description: DoR was defined only for patients who had an objective response, as the time in days from date of first documentation of response (CR/PR) until date of disease progression. CR was disappearance of all target lesions since baseline; any pathological lymph nodes selected as TL to have a reduction in short axis to <10 mm. At least a 30% decrease in the sum of the diameters of TL, taking as reference the baseline sum of diameters.
Time Frame: as for outcome 3
Population: Only patients in the ITT analysis set (which included all randomised patients), who also had an objective response and had measurable disease at baseline were included in the DoR analysis (n=89 for Fulvestrant arm and n=88 for Anastrozole arm).
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Fulvestrant 500 mg | Anastrozole 1 mg
Number analyzed (Participants) | 89 | 88
Months | 20.0 [10.6 to NA] — NA = Not Available. 75th percentile value not calculable due to insufficient data. | 13.2 [8.3 to 24.7]

5. Secondary Outcome: Expected Duration of Response (EDoR) for Fulvestrant Treatment Versus Anastrozole Treatment
Description: EDoR was estimated using the formula EDoR = p Efp(x), where x = DoR, p = proportion of responders, and Efp(x) = mean duration of response for responders. The estimation was completed by using the maximum likelihood estimates of p and Efp(x), as described by Ellis (Ellis S et al. Analysis of duration of response in oncology trials, Contemp Clin Trials 2008; 29:456-65).
Time Frame: Baseline RECIST 1.1 assessments and then every 12 weeks until disease progression or treatment discontinuation (up to approximately 38 months)
Population: EDoR analysis was based on the number of patients in the ITT analysis set (which included all randomised patients) who had measurable disease at baseline (n=193 for Fulvestrant arm and n=196 for Anastrozole arm).
Measure: Number; unit: Days
Arm/Group | Fulvestrant 500 mg | Anastrozole 1 mg
Number analyzed (Participants) | 193 | 196
Days | 346.84 | 227.58
Statistical Analysis 1: Comparison: Fulvestrant 500 mg vs Anastrozole 1 mg; Test type: Superiority or Other; p = 0.0367, Method of Ellis et al — 2-sided p-value; Rato of EDoR = 1.52, 95% CI 2-sided [1.03 to 2.26]

6. Secondary Outcome: Clinical Benefit Rate (CBR) for Fulvestrant Treatment Versus Anastrozole Treatment
Description: CBR was defined as the percentage of patients who had a clinical benefit (i.e. best objective response of CR, PR or stable disease), that was maintained for at least 24 weeks, prior to any evidence of progression. Note that a minimum duration of 22 weeks for CBR was applicable in the analysis (rather than 24 weeks) to allow for the protocolled window of +/-2 weeks.
Time Frame: as for outcome 3
Population: The ITT analysis set included all randomised patients.
Measure: Number; unit: Percentage of participants
Arm/Group | Fulvestrant 500 mg | Anastrozole 1 mg
Number analyzed (Participants) | 230 | 232
Percentage of participants | 78.3 | 74.1
Statistical Analysis 1: Comparison: Fulvestrant 500 mg vs Anastrozole 1 mg; Test type: Superiority or Other; p = 0.3045, Regression, Logistic — 2-sided p-value; Odds Ratio (OR) = 1.253, 95% CI 2-sided [0.815 to 1.932]

7. Secondary Outcome: Duration of Clinical Benefit (DoCB) for Fulvestrant Treatment Versus Anastrozole Treatment
Description: DoCB was defined only for patients who had clinical benefit, as the time in days from date of randomisation until the date of disease progression.
Time Frame: as for outcome 3
Population: Only patients in the ITT analysis set (which included all randomised patients) who also had a clinical benefit were included in the DoCB analysis (n=180 for Fulvestrant arm and n=172 for Anastrozole arm).
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Fulvestrant 500 mg | Anastrozole 1 mg
Number analyzed (Participants) | 180 | 172
Months | 22.1 [11.2 to NA] — 75th percentile value not calculable due to insufficient data. | 19.1 [11.3 to 30.4]

8. Secondary Outcome: Expected Duration of Clinical Benefit (EDoCB) for Fulvestrant Treatment Versus Anastrozole Treatment
Description: EDoCB was estimated using the formula EDoCB = p Efp(x), where x = EDoCB, p = proportion of responders, and Efp(x) = mean duration of response for responders. The estimation was completed by using the maximum likelihood estimates of p and Efp(x), as described by Ellis (Ellis S et al. Analysis of duration of response in oncology trials, Contemp Clin Trials 2008; 29:456-65).
Time Frame: as for outcome 3
Population: The ITT analysis set included all randomised patients.
Measure: Number; unit: Days
Arm/Group | Fulvestrant 500 mg | Anastrozole 1 mg
Number analyzed (Participants) | 230 | 232
Days | 667.94 | 532.04
Statistical Analysis 1: Comparison: Fulvestrant 500 mg vs Anastrozole 1 mg; Test type: Superiority or Other; p = 0.0561, Method of Ellis et al — 2-sided p-value; Ratio of EDoCB = 1.26, 95% CI [0.99 to 1.59]

9. Secondary Outcome: Comparison of the Effect of Fulvestrant Treatment Versus Anastrozole Treatment on Time to Deterioration of Health-Related Quality of Life (HRQoL)
Description: The Functional Assessment of Cancer Therapy - Breast (FACT-B) questionnaire was the instrument selected to assess HRQoL and comprised of following subscales: physical well-being (PWB), functional well-being (FWB), social well-being, emotional well-being, and breast cancer subscale (BCS). The main outcome measure from the FACT-B questionnaire was the Trial Outcome Index (TOI), which was a summary of the following subscales: PWB, FWB, and BCS. Outcome measure is reported as median time to deterioration, defined as the interval from the date of baseline of final analysis to the first assessment of worsened without an improvement in the next 12 weeks in FACT-B TOI, or the date of death (by any cause in the absence of symptom deterioration). Time to deterioration as measured by FACT-B total score was derived similarly and is also reported.
Time Frame: Quality of life questionnaires administered at 3 months post objective disease progression, then at 6-monthly intervals (approximately 75 months)
Population: The ITT analysis set included all randomised patients.
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Fulvestrant 500 mg | Anastrozole 1 mg
Number analyzed (Participants) | 230 | 232
months
  Time to TOI deterioration | 14.1 [5.5 to 44.1] | 11.1 [5.5 to 38.3]
  Time to FACT-B total score deterioration | 13.8 [5.5 to 38.7] | 11.1 [4.8 to 33.6]
Statistical Analysis 1: Comparison: Fulvestrant 500 mg vs Anastrozole 1 mg; Comparative statistical analysis for time to deterioration of TOI score is presented (fulvestrant versus anastrozole); Test type: Superiority or Other; p = 0.2846, Log Rank — 2-sided p-value; Stratified log-rank test with factors for prior chemotherapy for locally advanced/metastatic disease and measurable/non-measurable disease at baseline; Hazard Ratio (HR) = 0.88, 95% CI 2-sided [0.70 to 1.11] — A hazard ratio < 1 favours fulvestrant
Statistical Analysis 2: Comparison: Fulvestrant 500 mg vs Anastrozole 1 mg; Comparative statistical analysis for time to deterioration of FACT-B total score is presented (fulvestrant versus anastrozole); Test type: Superiority or Other; p = 0.0844, Log Rank — 2-sided p-value; [statistical method as in outcome 9, analysis 1]; Hazard Ratio (HR) = 0.82, 95% CI 2-sided [0.66 to 1.03] — A hazard ratio < 1 favours fulvestrant

ADVERSE EVENTS:
Time Frame: 116 months (duration from first patient enrolled to data cut-off for the final analysis)
Description: All-Cause Mortality: The ITT analysis set included all randomised patients. For serious adverse events and other (non-serious) adverse events: Safety population was defined as all patients who received at least 1 dose of randomised study medication. 2 patients in the Fulvestrant 500 mg arm did not receive treatment and were not included in the safety population.
Arm/Group | Fulvestrant 500 mg | Anastrozole 1 mg
All-Cause Mortality (participants affected / at risk) | 157/230 | 159/232
Serious Adverse Events (participants affected / at risk) | 39/228 | 36/232
Other Adverse Events (participants affected / at risk) | 125/228 | 127/232
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fulvestrant 500 mg (N=228) | Anastrozole 1 mg (N=232)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 2 (6)
Anaemia macrocytic (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Jaundice cholestatic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 2 (2)
Device related sepsis (Infections and infestations) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 2 (2)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Peritonitis (Infections and infestations) | 2 (2) | 0 (0)
Pneumonia (Infections and infestations) | 3 (3) | 4 (7)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 3 (3)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Traumatic spinal cord compression (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Hepatic enzyme increased (Investigations) | 0 (0) | 1 (2)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Acoustic neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma of the oral cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Brain oedema (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 2 (2) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 2 (2)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 7 (10) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 1 (1)
Circulatory collapse (Vascular disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 2 (2)
Hypertensive crisis (Vascular disorders) | 2 (2) | 0 (0)
Duodenal stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large intestine perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal dilatation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fulvestrant 500 mg (N=228) | Anastrozole 1 mg (N=232)
Anaemia (Blood and lymphatic system disorders) | 9 (10) | 20 (21)
Cough (Respiratory, thoracic and mediastinal disorders) | 12 (15) | 9 (12)
Fatigue (General disorders) | 29 (35) | 18 (20)
Injection site pain (General disorders) | 12 (15) | 10 (23)
Oedema peripheral (General disorders) | 11 (11) | 14 (15)
Alanine aminotransferase increased (Investigations) | 16 (18) | 8 (8)
Aspartate aminotransferase increased (Investigations) | 12 (13) | 9 (9)
Arthralgia (Musculoskeletal and connective tissue disorders) | 42 (65) | 31 (40)
Back pain (Musculoskeletal and connective tissue disorders) | 22 (25) | 18 (19)
Myalgia (Musculoskeletal and connective tissue disorders) | 16 (19) | 8 (11)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 17 (22) | 11 (15)
Headache (Nervous system disorders) | 12 (13) | 12 (12)
Anxiety (Psychiatric disorders) | 12 (13) | 4 (4)
Insomnia (Psychiatric disorders) | 18 (19) | 15 (16)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 15 (17)
Hot flush (Vascular disorders) | 26 (35) | 24 (32)
Hypertension (Vascular disorders) | 18 (19) | 22 (25)
Constipation (Gastrointestinal disorders) | 16 (16) | 11 (13)
Diarrhoea (Gastrointestinal disorders) | 15 (20) | 15 (17)
Nausea (Gastrointestinal disorders) | 25 (29) | 25 (27)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-12-17): https://cdn.clinicaltrials.gov/large-docs/80/NCT01602380/Prot_000.pdf
  • Statistical Analysis Plan (2022-05-03): https://cdn.clinicaltrials.gov/large-docs/80/NCT01602380/SAP_001.pdf